CLINICAL TRIAL: NCT04059211
Title: Sensitivity and Specificity of Urinary Dipstick in Emergency Departments
Status: Completed | Type: Observational
Sponsor: Sonderborg Hospital (Other Government)
Responsible Party: Principal Investigator, Jan Dominik Kampmann, Medical doctor, Sonderborg Hospital
Other Study IDs: S-20190013
Record Dates: First submitted 2019-08-15; First posted 2019-08-16 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Proteinuria
Keywords: urinary dipstick; emergency department
MeSH Terms: conditions — Proteinuria; Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Urinary dipstick — Sensitivity and specificity of urinary dipstick for proteinuria in emergency departments

SUMMARY:
Urinary dipsticks are commonly used in emergency departments since they are a cheap and quick diagnostic tool. However the sensitivity and specificity of urinary dipsticks might be compromised in emergency departments due to fluid imbalance and acute illness itself.

DETAILED DESCRIPTION:
The study is designed as a prospective observational study on the emergency department in Sonderborg, Southern Denmark.

All patients above 18 years of age who have given their consent are included. Urinary dipstick and albumin creatinine ratio is obtained simultaneously within 48 hours after admission on the emergency department.

Patient with a positive urinary dipstick will be asked to deliver another urinary dipstick and albumin creatinine ratio 3-8 weeks later.

To our knowledge has the specificity and sensitivity of urinary dipstick for protein not been described, yet. Our design will give us the possibility not only to quantify specificity and sensitivity in the acute phase on the emergency department but in the non-acute phase after discharge from the emergency department, as well.

ELIGIBILITY:
Inclusion Criteria:

* All patients above 18 years of age who were admitted to the emergency department in Sonderborg and who gave their consent

Exclusion Criteria:

* anuria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients above 18 years of age who were admitted to the emergency department in Sonderborg and who gave their consent.
Sampling Method: Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of urinary dipstick for proteinuria on emergency departments | 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sonderborg Hospital, Sønderborg, Southern Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided